CLINICAL TRIAL: NCT05858268
Title: The NeuralNET: Research to Impact Diagnosis, Mechanistic Understanding and Treatment of Children's Brain and Mental Health Disorders - A Pilot Study in Cerebral Palsy
Brief Title: NeuralNET Cerebral Palsy Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Rosetrees Trust (Other); Isaac Newton Trust (Unknown); National Institute for Health Research, United Kingdom (Other Government); Illumina, Inc. (Industry)
Responsible Party: Principal Investigator, Heather Pierce, Research Study Coordinator, University of Cambridge
Other Study IDs: IRAS: 319781
Record Dates: First submitted 2023-04-24; First posted 2023-05-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Whole-genome sequencing — Whole-genome sequencing

SUMMARY:
The NeuralNET Cerebral Palsy Pilot Study is testing a genetic testing pathway in the NHS for children with cerebral palsy (CP). Other studies suggest that almost one in three peoples' CP is caused by a change in their genes, but more studies are needed to confirm this. A genetic test called whole genome sequencing (WGS) will be used for children who have CP to look for rare changes in genes that cause the condition, and the results of the test will be given to children's doctors within 12 weeks. Knowing that CP has a genetic cause could lead to changes being made to a child's care or treatment that could improve their condition.

The study will test 66 children with CP from 3 hospitals, and also their biological parent(s), if they're available. Following informed consent, the investigators will collect a blood sample from everyone taking part which will be sent for WGS. It is important to understand what families think and feel about the testing. The investigators will ask parents/guardians of the children taking part to fill in two questionnaires, one before and one after WGS. Some parents/guardians will also be interviewed after getting the WGS result, to ask about their experience of the testing. The study will take up to 16 months per family.

The results of this pilot study will tell the investigators if it is feasible for the NHS to use WGS to test children with CP. If so, a larger study testing more children with CP can then be carried out to help decide if this type of WGS-based testing should be made available through the NHS to children with CP whose clinical care might be changed by the result. The genetic findings from this study will also be made available to other researchers and doctors to do more research into CP that might help improve general understanding of the condition and its potential treatment.

ELIGIBILITY:
Inclusion Criteria:

Children with cerebral palsy (CP):

1. Has a clinical diagnosis of CP in the medical record
2. Any GMFCS score (GMFCS 1-5)
3. Does not have a known genetic diagnosis that explains the CP phenotype
4. Has a parent/legal guardian available who can consent and is willing to complete study questionnaires
5. Invited to participate by a clinician at a participating recruitment site

Biological parents of children with CP will also be included in the study if they are:

1. A biological parent of the child
2. Aged 18 years or above
3. Willing and able to give informed consent for participation in the study Participant type

Exclusion Criteria:

Children with cerebral palsy (CP):

1. Children that have a pre-existing genetic diagnosis from whole genome sequencing or whole-exome sequencing
2. Children not matching the inclusion criteria

Biological parents of children with CP will be excluded from the study if they do not meet the biological parent inclusion criteria i.e. they ARE NOT:

1. A biological parent of the child
2. Aged 18 years or above
3. Willing and able to give informed consent for participation in the study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a clinical diagnosis of cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of rapid whole-genome sequencing of children with cerebral palsy | 16 months
  The investigators will measure feasibility of rapid whole-genome sequencing of children with cerebral palsy by successful delivery of WGS results to 66 children with a clinical diagnosis of CP within 12 weeks of blood sample receipt in the laboratory.

SECONDARY OUTCOMES:
Uptake of WGS testing by families with a child with CP | Baseline
  The percentage of uptake of WGS testing by families with a child with CP will be measured by comparing the number of families invited to the study to the number who proceed with testing at baseline
Reasons for declining offer of WGS | 16 months
  The reasons for declining the offer of WGS provided by families voluntarily to the referring clinician will be measured in aggregate using a questionnaire at the close of the recruitment
Identification of specific genetic contributors to CP in the UK | 16 months
  Specific genetic contributors to CP in children in the UK will be measured using the collation of WGS results at the close of the recruitment
Parent/guardian intolerance for uncertainty | baseline
  Intolerance of uncertainty of parent/guardian will be measured with the short version of the validated Intolerance for Uncertainty scale, which is a 12-item self-administered questionnaire where items are rated on a 5-point Likert scale where a higher score means higher intolerance of uncertainty.
Parent/guardian attitude to genome sequencing | baseline and 16 months
  Four-item scale via self-administered questionnaire examining general attitudes (eg harmful vs. beneficial, unimportant vs. important, etc.) of parent/guardian to genome sequencing measured on a five-point Likert scale, where a higher score means more positive attitude.
Parent/guardian decisional conflict | baseline
  Parent/guardian decisional conflict will be measured with validated sixteen-item self-administered questionnaire which assesses decisional certainty or conflict about a healthcare decision on a five-point Likert scale, where a higher score indicates higher uncertainty or conflict.
Parent/guardian empowerment | baseline, 16 months
  Parent/guardian empowerment relating to genomic medicine will be measured with the Genomics Outcome Scale, a validated six-item self-administered questionnaire with a 5-point Likert scale, where a higher score indicates higher theoretical construct of empowerment.
Parent/guardian decisional regret | 16 months
  Parent/guardian decisional regret about WGS will be measured with a validated 5-item self-administered Decisional Regret Scale, which uses a 5-point Likert scale where higher scores indicate greater decisional regret.
Parent/guardian psychological impact of WGS | 16 months
  Parent/guardian psychological impact of WGS will be measured with adapted 10-item version of the validated Feelings About genomic Testing Results (FACToR) scale, which uses a 5-point Likert scale to measure agreement with specific feelings about the impact of result disclosure after genomic testing, where a higher score indicates greater agreement with those feelings.
Impact of WGS on family quality of life | 16 months
  Impact of WGS on the family's quality of life will be measured using the Family Impact Module of The PEDS-QL, which is a 36-item validated self-administered scale. It uses a 5-point Likert scale where higher scores indicated greater agreement with specific items.
Clinical utility of WGS testing in children with CP | 16 months
  The clinical utility of WGS testing in children with CP from the Paediatrician's perspective will measured using the validated Clinician-reported Genetic testing Utility InDEx (C-GUIDE), a self-administered questionnaire which includes 17 items related to results received for the primary indication for testing and 9 items related to secondary variant results received. Individual items scores range from -1 to 2. An item score >0 indicates positive utility, item scores <0 indicate presence of negative utility, and item scores of 0 indicate absence of utility.
Number of candidate variants which warrant further investigation of pathogenicity | 16 months
  Number of candidate variants which warrant further investigation of pathogenicity via collaborative studies will be measured by collating potentially pathogenic variants of uncertain significance at the completion of the study.
Generation of data to support the refinement of clinical criteria for WGS for CP | 16 months
  Data to support the refinement of clinical criteria for assessing CP patient suitability for WGS testing will be measured using the correlation of clinical features with identification of causative variants by WGS

CONTACTS AND LOCATIONS:
Overall Officials: David Rowitch, MD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://www.eastgenomics.nhs.uk/research/neural-net-research-project/